CLINICAL TRIAL: NCT00710489
Title: Potential Research Study Participant Registry
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 287381
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Acne; Actinic Keratosis; Dysplastic Nevi; Eczema; Psoriasis; Skin Cancer; Rosacea; Leg Ulcers; Foot Ulcers; Atopic Dermatitis
Keywords: Acne; Actinic Keratosis; Dysplastic Nevi; Eczema; Psoriasis; Vitiligo; Skin Cancer; Rosacea; Leg or Foot Ulcers; Atopic Dermatosis
MeSH Terms: conditions — Acne Vulgaris; Keratosis, Actinic; Dysplastic Nevus Syndrome; Eczema; Psoriasis; Skin Neoplasms; Rosacea; Leg Ulcer; Foot Ulcer; Dermatitis, Atopic; Vitiligo

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the potential research study participant registry is to keep potential research subjects informed about any future research studies in which they may meet the criteria for enrollment. The purpose of this study is also to assist current and future clinical trials with recruitment of subjects.

DETAILED DESCRIPTION:
Methods:

Subjects will self identify themselves via the UCDMC Dermatology website to complete a survey regarding their interest in learning about future dermatology clinical research projects. Subjects provide contact information and check of a list of potential topics of interest.

Procedures:

Potential participants will find a link on the UCDMC Dermatology website to our registry. The potential participant will read information about the registry. If they wish additional information, they can follow a link to the potential research registry consent form. At this stage, the potential participant may answer, "no" to the consent form and they will be redirected back to the Clinical trials website. If they answer, "yes" then they will be linked to the registry questionnaire. The potential subject would then decide if they want to participate in the registry and if so what information they want to provide. The Clinical Research Coordinators would contact potential study participants to see if they meet the eligibility criteria for any of our current studies.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult community members with an interest in one or more of the following dermatologic conditions: Acne, Actinic Keratosis, Blistering Diseases, Dysplastic Nevi (mole), Eczema, Psoriasis, Vitaligo, Skin Cancer Prevention, Skin Cancer Treatment, Phototherapy Treatment Options, Rosacea, Leg or Foot Ulcers, Lichen Planus, Atopic Dermatosis, Canker Sores,others as indicated.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2008-05; Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Identify Dermatology Clinical research topics of interest in the community. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tong Liu, M.D., Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical